CLINICAL TRIAL: NCT05856968
Title: To Investigate the Effect of Continuous Versus Interrupted Subcutaneous Fat Closure in Reducing Surgical Site Infection Among Over-weight or Obese Women Who Are Undergoing Elective Caesarean Section
Brief Title: Investigation of Continuous Versus Interrupted Subcutaneous Fat Closure in Reducing Surgical Site Infection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of The West Indies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CREC-MN.0296,2021/2022
Record Dates: First submitted 2023-05-03; First posted 2023-05-12 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy, Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Doctors at the Victoria Jubilee hospital will perform continuous or interrupted subcutaneous tissue closure resulting in the reduction of the occurrence of surgical site infection on overweight and obese women
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- continuous subcutaneous tissue closure (Active Comparator): continuous subcutaneous tissue closure
  Interventions: Procedure: continuous subcutaneous tissue closure
- Interrupted subcutaneous tissue closure (Active Comparator): Interrupted subcutaneous tissue closure
  Interventions: Procedure: Interrupted subcutaneous tissue closure

INTERVENTIONS:
Procedure: continuous subcutaneous tissue closure — The use of continuous subcutaneous tissue closure to determine which closure results in a lower rate of surgical site infection.
  Arms: continuous subcutaneous tissue closure
Procedure: Interrupted subcutaneous tissue closure — The use of interrupted subcutaneous tissue closure to determine which closure results in a lower rate of surgical site infection.
  Arms: Interrupted subcutaneous tissue closure

SUMMARY:
This research aims to clarify the best way to perform subcutaneous tissue closure in overweight and obese patients undergoing caesarean section to reduce the occurrence of surgical site infections. This Study seeks to get some local perspective on the need for and type of subcutaneous fat closure in obese women undergoing cesarean section, thereby reducing Surgical Site Infection. This is a pilot; double- blinded randomized control trial, with balanced randomization (1:1) and parallel grouped study. The sample size calculated by Raosoft Sample Size Calculator Software determined that based on a margin of error of 5%, there would need to be 266 participants to give 90% confidence level to detect a significant difference between both arms of the study. Patients who are immune-compromised, those with anemia, requiring transfusion will be excluded from the study, also any mother who wishes not to participate. Patients will be reviewed 7 days post operatively. Wound complications will be identified by a questionnaire by telephone at 4 weeks and 3 months post operatively. Data will be collected from Specific closed answer questions. Data extraction sheet will be used to collect data for the patient. This information will be collected either from the docket, direct review or examination of the study participants. The research will be done at Victoria Jubilee Hospital. The Research will last six months.

DETAILED DESCRIPTION:
Background and Rationale for the study

Caesarean Section is the most common abdominal operation performed worldwide. At the Victoria Jubilee Hospital, the C-Section rate is 23.2% for 2021. Wound complications are encountered in about 3-15% (5) of women undergoing C- section and this includes: hematomas, seromas and wound infections. Given the trend of rising C-Section rate, the associated complications also increase. Obesity has a direct effect on wound complication rate. Obesity is a complex medical disorder characterized by an excess of total body fat. A body max index (BMI) of 25 kg/m2 to < 30 kg/m2 constitutes overweight and obesity with a BMI of 30 kg/m2.Data from the 2016/17 Jamaica Health and Lifestyle Survey showed that one in two Jamaicans or 54% were overweight or obese. The data further revealed that women are more affected by overweight/obesity, with two-thirds of Jamaican women 15 years or older being overweight or obese (4).

Abdominal wall closure is performed traditionally by using a 3 layer technique in which the parietal peritoneum with the posterior rectus sheath, anterior rectus sheath and skin are individually and sequentially closed. Camper's fascia provides a potential space for hematoma and seroma formation. The vascular supply to subcutaneous fat is relatively poor making the tissue susceptible to infection. A good surgical technique is the one that eliminates the dead space in subcutaneous tissue and approximates edges without tension. The suturing of subcutaneous tissue aims to reduce the risk of formation of fluid reservoirs theoretically reducing the rate of postoperative hematoma and seroma development.

A Meta-Analysis of 6 studies showed that suturing reduces the risk of wound complications by 34% in subcutaneous tissue greater than 2cm. Only a small number of research studies evaluated the impact of various subcutaneous tissue closure methods at C-Section (1).

A Retrospetive study between 2008 to 2018 compared surgical site infections (SSI) between continuous versus interrupted subcutaneous tissue closure during cesarean delivery in women with fat thickness > 2cm. The study concluded that continuous subcutaneous tissue closure yielded a lower rate of surgical site infection complications compared to interrupted subcutaneous tissue closure (2).

A Randomized controlled trial was done in Egypt March 2018 among obese women undergoing cesarean delivery. This study concluded that most surgical wound complications were reduced if continuous subcuticular sutures were replaced with interrupted one (1).

It was further noted that the above studies were conducted internationally. We therefore saw the need for a similar study locally to test these international findings in a socially and culturally divergent population. Hopefully this study will provoke further studies which may eventually influence the management strategies employed at VH and other local hospitals in the prevention of SSI. Given the high numbers of Cesarean Sections performed worldwide and locally, any preventive measures that could possibly help reduce the incidence of wound complications would

Aims and Objectives

This research aims to further clarify the best way to perform subcutaneous tissue closure in our overweight and obese patients undergoing caesarean section so as to reduce the occurrence of surgical site wound infections.

Doctors at the Victoria Jubilee hospital will perform continuous or interrupted subcutaneous tissue closure resulting in the reduction of the occurrence of surgical site infection on overweight and obese women between September 2025 and September 2026.

The objective is to determine which method of subcuticular closure is superior at reducing surgical site infections in obese women undergoing cesarean section.

The objective includes:

* Providing and improving knowledge of use and benefit of subcuticular suturing in obese women undergoing cesarean section.
* Determining the effectiveness of one subcuticular suture technique over another in reducing Surgical Site Infection

Main Hypothesis: The use of continuous subcuticular closure is superior to interrupted closure in reducing SSI in obese women undergoing cesarean section.

Hypothesis 0: There is no difference in reducing SSI based on suture techniques Hypothesis 1: The occurrence of SSI is reduced in the continuous suture technique group

Methodological Design

Overall Study Design (Theoretical Framework):

This Study is a pilot; double- blinded randomized control trial, with balanced randomization (1:1) and parallel grouped study.

The obese/overweight patient will be selected from the booking Antenatal Clinic (ANC) at the Victoria Jubilee Hospital. They will be sensitized by the nurse in charge and also fliers advertizing the study to be embarked upon. The nurse will be sensitized about the inclusion criteria for these patients to partake in the study. The participants who wish to partake in the study, their record will be colour coded. There will be a master list of all participants partaking in the study. The patients will be equally randomized to either arm of the study by a computer generated random allocation sequence to ensure allocation concealment into two groups. The allocation sequence will be concealed from the researcher enrolling and assessing participants in sequentially numbered order listing. Determination of a participant to 1 of 2 treatment groups will be made by reference to a statistical series based on random sampling by a chosen resident. The details of the series will be unknown to any of the investigators or to the co-ordinator of the study. The resident will have a master list with the participant´s name who will be randomly selected and placed In an arm of the study already. Patients and Physicians will be blinded after the assignment of each arm of intervention. Data Collectors will also be unaware of which arm of the study each participant is attached. All randomized participants will be used in the analysis and retained in the group to which they will be allocated. The intention to treat analysis will be used to preserve the benefit of randomization. The primary analysis will be intention to treat and involve all patients who are randomly assigned.

Location and Time Frame of the study Victoria Jubilee Hospital: Antenatal Clinic and Labour Ward will be used for patient selection as these places would be where the Antenatal patients have their first encounter with the institution. Institutional approval from South East Regional Authority would be required.

Research Procedures/Protocols - Data Collection/Research Intervention Procedures

There will be a metre stick, tape measure or height measuring scales used to document height of participants in metres.

Existing scales will be used to measure the weight in kg, to complete calculation of BMI.

Specific closed answer questions regarding the incision site will be asked to assess any thought of SSI when patients are reviewed Patients will be randomly recruited from the Antenatal clinic. The docket will be colour coded for each participant of the study.

The surgeon at the time of surgery will be informed of the type of subcuticular suturing to be done. This will already be randomized from the masters list previously.

The proposed suture for subcuticular closure will be 1 vicryl round bodied and skin closure will be 2/0 prolene. The use of a stat dose of ceftriaxone will be used for all patients participating in the study.

They will be informed of the process of their surgery and any possible complications, including Surgical Site Infection.

The Patient will be required to sign an informed consent form giving permission.

The Wards and the operation theatre will be sensitized about the Study with laminated posters/flyers.

These patients will be reviewed on Day 3 post-operatively on the surgical ward. The patients will also be reviewed on Day 7. During Week 4 and Week 12 post-operatively they will be reviewed via a telephone conversation and asked specific closed answer questions regarding the incision site to assess any thought of SSI when being reviewed. Confidentiality will be maintained by securing these questionnaires in a locker that will have a numbered lock on the ward or records office.

If a patient is discovered to have a SSI, they will be advised to visit the ward and an assessment made of the severity. These patients will be treated with culture directed antibiotics and daily dressing or alternate day dressing until the SSI has resolved.

Data extraction sheet will be used to collect data for the patient. This information will be collected either from the docket, direct review or examination of the study participants. A spreadsheet table will have parameters such as Study ID number, Demographics, Preoperative medication, Indication for C- Section, type of abdominal incision, type of subcutaneous closure, blood loss (intraoperative event), Length of surgery and Type of suture for skin closure.

Methods of Data Analysis The data will be analyzed using the appropriate statistical test from STATA version 11.2. Descriptive Analysis, Chi-Square analysis and other appropriate analyses of association will be used to analyze the data. A sample size of 266 patients will be assessed, 133 patients for each group.

Methods for storing and securing study/biological data The research information will be stored in a secured, fire-proof filing cabinet. The computer used for the spreadsheet parameters will be password protected and logged off when not in use.

Methods for protecting participants' confidentiality The Patients´ name will not be used and only study ID numbers from medical records will be available as a way to trace these patients. Questionnaires will be secured in a number- maintained locker in the records office. There will also be a master list linking the study ID to the participant´s medical records number that will be stored confidentially and separately.

Indicate what is the level of risk associated with this research

No more than minimal risk

Please describe risk, discomfort (physical/psychological), inconvenience, side effects, and financial costs to participants (include measures to mitigate these risks/discomforts)

Nil Physical discomfort Nil inconvenience/side effects, seeing that these are already interventions that are commonly employed to closing subcutaneous tissues in obese patients.

Indicate direct benefits to participants This may reduce the risk of developing a surgical site infection post- operatively in obese women (1); while determining which closure is superior at reducing SSI.

Impacts of the study on human groups that are not participants in the study (positive/negative, where applicable) The impact of this study may lead to protocols being implemented for obese/ overweight patients undergoing Cesarean Section so as to reduce the risk of SSI.

Describe process for informed consent.

There will be a resident in the booking clinic at VJH who will be consenting the participants in this study. This resident will not be a member of the clinical managing team. One method of closure is being tested against the other as a way of reducing SSI will be advised to these participants. They will be sensitized about the various stages/ types of SSI that may arise and method of treatment to be used if there is an occurrence.

How the results will be disseminated?

A report will be produced and possibly implemented within the protocols of Cesarean Delivery for Overweight/Obese patients

How the results will be acted upon for both the participants and the community?

The impact of this study should lead to protocols being implemented in these obese/overweight patients undergoing C Section and adapted by the infection control committee to reduce the incidence of SSI.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/Obese Women > 25kg/m2, measured in the first trimester
* Single Fetus
* Gestational Age (37-41) week calculated by sure dates and confirmed by first trimester ultrasound
* Elective Lower Segment Cesarean Section

Exclusion Criteria:

* Patients who are immune-compromised e.g. Known Diabetes Mellitus or HIV positive mothers
* Patients who are on long term Steroid use: e.g. SLE, Rheumatoid Arthritis
* Multifetal Pregnancy
* Those with anemia, requiring transfusion
* Obstetric Complications: e.g. Placenta Previa
* Any mother who wishes not to participate in the study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Surgical Site infection | 12 weeks
  Patients will be reviewed on Day 3 post-operatively on the surgical ward. The patients will also be reviewed on Day 7. During Week 4 and Week 12 post-operatively they will be reviewed via a telephone conversation and asked specific closed answer questions regarding the incision site to assess any thought of SSI when being reviewed.

REFERENCES:
- [Background] Alalfy M, Elgazzar A, Fares T, Nagy O, Ellithy A, Lasheen Y, Kamel A, Soliman M, Hassan A, Samy A, Taher AM, Ogila AI, Saad H, Salah H, Ramadan M, Nabil M, Hatem DL, Fikry M. Effect of subcutaneous tissue closure technique in cesarean section on postoperative wound complications in obese Egyptian women. J Matern Fetal Neonatal Med. 2019 Aug;32(15):2452-2459. doi: 10.1080/14767058.2018.1438399. Epub 2018 Feb 20. PMID 29415592
- [Background] Lauterbach R, Ben David C, Bachar G, Justman N, Matanes E, Ginsberg Y, Vitner D, Beloosesky R, Weiner Z, Zipori Y. Continuous versus disrupted subcutaneous tissue closure in cesarean section: A retrospective cohort study. Int J Gynaecol Obstet. 2023 Jan;160(1):113-119. doi: 10.1002/ijgo.14322. Epub 2022 Jul 15. PMID 35766992
- [Background] Caribbean Institute for Health Research (CAIHR) (JA) Jamaica Health and Lifestyle Survey III (2016- 2017). Available from: https://www.moh.gov.jm/wp-content/uploads/2018/09/Jamaica-Health-and-Lifestyle-Survey-III-2016-2017.pdf
- [Background] Zuarez-Easton S, Zafran N, Garmi G, Salim R. Postcesarean wound infection: prevalence, impact, prevention, and management challenges. Int J Womens Health. 2017 Feb 17;9:81-88. doi: 10.2147/IJWH.S98876. eCollection 2017. PMID 28255256